CLINICAL TRIAL: NCT04032119
Title: Multicenter Randomized Controlled Trial of Gastric Endoscopic Submucosal Dissection With or Without Epineprhine Added Solution
Brief Title: RCT of Gastric ESD With or Without Epineprhine Added Solution
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Osaka International Cancer Institute (Unknown); Fukuoka University (Other); Changi General Hospital (Other); Kyoto 2nd Red Cross Hospital (Unknown); Ishikawa Prefectural Central Hospital (Unknown); Kosin University Gospel Hospital (Other); Machida General Hospital (Unknown); Nara City Hospital (Unknown); Wakayama Red Cross Hospital (Unknown); JCHO Osaka Hospital (Unknown); Sapporo Kinentou hospital (Unknown); Japan Community Healthcare Organization Osaka Hospital (Unknown)
Responsible Party: Principal Investigator, Hon Chi Yip, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EPI-ESD RCT01
Record Dates: First submitted 2019-07-23; First posted 2019-07-25 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Gastric Neoplasm; Early Gastric Cancer
Keywords: Gastric Endoscopic submucosal dissection; Epinephrine
MeSH Terms: conditions — Stomach Neoplasms | interventions — Endoscopic Mucosal Resection; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Epinephrine (Experimental): 0.2ml 1:10000 epinephrine diluted into each 20ml of the original solution for submucosal injection
  Interventions: Procedure: Endoscopic submucosal dissection; Drug: Epinephrine
- Non-epinephrine (Active Comparator): No epinephrine would be added into the solution
  Interventions: Procedure: Endoscopic submucosal dissection

INTERVENTIONS:
Procedure: Endoscopic submucosal dissection — Endoscopic submucosal dissection
Drug: Epinephrine — Epinephrine
  Arms: Epinephrine

SUMMARY:
This is an international multi-center randomised controlled study comparing outcomes of gastric endoscopic submucosal dissection (ESD) with or without addition of epinephrine in the submucosal injection solution.

DETAILED DESCRIPTION:
Endoscopic submucosal dissection (ESD) is an endoscopic technique aiming to achieve en-bloc resection of mucosal neoplastic lesion in the gastrointestinal tract. It is now considered as the standard of treatment for early gastric cancer confined to the mucosa, achieving an excellent overall survival comparable to that of surgical resection.

Important adverse events associated with gastric ESD include hemorrhage (intraoperative or delayed) and perforation. The reported incidence of intraprocedural and delayed hemorrhage of gastric ESD is generally higher than that of esophageal or colorectal ESD5. This is likely due to the rich blood supply of the stomach penetrating from the muscularis to the submucosal layer. Bleeding during ESD would result in difficulty in visualizing the correct plane of dissection from blood clots obscuring view of the endoscope. As a result, prolonged procedural time may be required to achieve hemostasis and obtain adequate view for dissection.

There are currently different options of the solution for submucosal injection during gastric ESD. Epineprhine has often been added into these solutions with the aim of causing vasoconstrictive effect and potentially reduce bleeding during the procedure. The use of epinephrine has been recommended when removing larger pedunculated polyps with endoscopic mucosal resection (EMR)6. However the exact clinical benefit of adding epinephrine during gastric ESD has not been proven in the literature. On the other hand, when larger dose of epinephrine is absorbed systemically it may rarely cause significant tachycardia and generalized vasoconstriction, putting patients at risk of myocardial infarction or cerebrovascular accident.

A retrospective propensity score analysis was previously performed in one of our Japanese center (Presented at JGCA 2019, Shizuoka). After adjustment of important confounding factors including age, sex, tumor location, specimen size, depth of tumor invasion, presence of histological ulcer or scar and operators' experience, the addition of epinephrine into submucosal solution was associated with a significantly shorter procedural time upon multivariate analysis. The mean procedural time was 72±54 minutes versus 93±62 minutes with and without epinephrine respectively. (p<0.001) With the encouraging result from a single center retrospective study, we plan to conduct a prospective multicenter randomized controlled study to confirm the benefit of adding epinephrine into the submucosal solution during gastric ESD.

ELIGIBILITY:
Inclusion Criteria:

* Selection criteria: Presence of intramucosal neoplastic lesions in the stomach planning for endoscopic submucosal dissection (Vienna Classification Category 3 and 4 lesion)
* Target subjects receiving sufficient briefing from the attending physician regarding the content of this study and providing informed consent for participation

Exclusion Criteria:

* Recurrent / remnant lesion after previous endoscopic resection
* Lesions arising from surgical anastomotic site, such as gastrojejunostomy / gastroduodenostomy.
* Marked electrolyte abnormalities
* Hemostatic or coagulative abnormalities
* Patient on anti-coagulant agents, including warfarin and other direct oral anti-coagulants (those on antiplatelet can be included)
* Failure of vital organ (heart, lungs, liver, or kidneys) function
* Allergic to components of injection solutions: Epinephrine, hyaluronic acid etc
* Other cases deemed by the examining physician as unsuitable for safe treatment

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Overall procedural time | During the endoscopic procedure
  From the beginning of mucosal incision till the end of submucosal dissection, excluding time for prophylactic homeostasis

SECONDARY OUTCOMES:
Number of intra-procedural hemorrhage events | During the endoscopic procedure
  The number of oozing or spurting bleeding events during a procedure, requiring hemostasis with coagulating forceps
Maximum systolic blood pressure | During the endoscopic procedure
  Maximum systolic blood pressure during ESD
Maximum heart rate | During the endoscopic procedure
  Maximum heart rate during ESD
Adverse event - Delayed hemorrhage | 30 days
  Delayed hemorrhage (Based on CTCAE definition)
Adverse event - Perforation | 30 days
  Perforation (Based on CTCAE definition)
Adverse event - Cardiovascular event | 30 days
  Cardiovascular event (Based on CTCAE definition)
Adverse event - Cerebrovascular event | 30 days
  Cerebrovascular event (Based on CTCAE definition)
Other adverse event | 30 days
  Based on CTCAE definition
Pathology | During the endoscopic procedure
  Final histology based on Vienna Classification
Size of lesion | During the endoscopic procedure
  Size of lesion
Depth of invasion | During the endoscopic procedure
  Depth of tumor invasion
Vertical margin | During the endoscopic procedure
  Vertical margin involvement
Horizontal margin | During the endoscopic procedure
  Horizontal margin involvement
Differentiation | During the endoscopic procedure
  Degree of differentiation for cancer of stomach
Lymphovascular invasion | During the endoscopic procedure
  Lymphovascular invasion on pathology

CONTACTS AND LOCATIONS:
Overall Officials: Hon Chi Yip, MBChB, FRCSEd, Principal Investigator — Chinese University of Hong Kong
Locations (7):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong
- Japan (4):
  - Ishikawa Prefecture Central Hospital, Ishikawa
  - Kyoto 2nd Red Cross Hospital, Kyoto
  - Osaka International Cancer Institute, Osaka
  - Shizuoka Cancer Center, Shizuoka
- Changi General Hospital, Singapore, Singapore
- Kosin University Gospel Hospital, Busan, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yip HC, Uedo N, Iwagami H, Waki K, Ohtsu K, Miyaoka M, Yao K, Akamatsu T, Konishi T, Nakano S, Nakanishi H, Doyama H, Machida H, Jung K, Chiu P, Iwasaki T, Uchita K, Kawamura T, Takizawa K, Kitamura Y, Li JW, Ang TL, Shimokawa T, Zhu Z, Yung MY. The use of diluted epinephrine during gastric endoscopic submucosal dissection: an international randomized controlled trial. Gastrointest Endosc. 2026 Jan 29:S0016-5107(26)00072-6. doi: 10.1016/j.gie.2026.01.031. Online ahead of print. PMID 41620139